CLINICAL TRIAL: NCT05950451
Title: Self-management Education in Multi-professional Health Centres
Acronym: ETHOPEE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC22_UF9821_ETHOPEE
Record Dates: First submitted 2023-07-11; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Self-management
Keywords: Patient education as topic; Primary health care; multimorbidity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention is led during this descriptive study

SUMMARY:
The goal of this observational study is to learn about the best educative and organizational dimensions favouring the development of self-management education in multiprofessional health centres. The main question is to identify the favorable characteristics in creation, implementation and maintenance in developing self-management education programme in multiprofessional health centres.

DETAILED DESCRIPTION:
The study wil be composed of 2 phases. Phase 1 will consist of a national questionnaire survey of French Regional Health Authorities (ARS) to identify and characterize all multiprofessional health centres running a self-management programme in France. It will be supported by the informal inter-ARS network of self-management project managers.

Phase 2 will consist of a qualitative survey of multiprofessional health centres. On the basis of the various significant variables identified in phase 1, different multiprofessional health centres will be selected to provide a varied sample (location, number of healthcare professionals, themes, etc.). This will enable an in-depth analysis of the findings of the quantitative survey, and a comparison with the realities of the multiprofessional health centre's health care professionals.

ELIGIBILITY:
First phase (quantitative survey): All regional health authority agencies will be surveyed on all self-management programmes developed by multiprofessional health centres since 2014 (estimated number of 270 in France in 2021).

Second phase (qualitative survey): In the first time, for the selection of the multiprofessional health centres , we will realized a varied sampling in search of maximum variation of the multiprofessional health centres according to the results of the first phase (continuation or not of the program, location of the programme, number of health care professionals in the educational team and presence of expert patients, theme of the programme...). In a second phase, for the individual interviews, we will carry out a varied sampling in search of maximum variation reflecting the plurality of the educational team observed in the documentary survey of each multiprofessional health centres.

The educational team includes healthcare professionals from the multiprofessional health centres and expert patients.

There is no exclusion criteria.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: For the first phase, the population study will be composed of all the regional health authorities agencies.
  For the second phase, the population study will be composed of 10 to 15 multiprofessional health centres, with in each 5 to 7 individual interviews with health care professionals. The population will be composed of 105 health care professionals
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Favourable educational and organizational dimensions to self-management in multiprofessional health centre | 9 months
  The outcome will consist of a description and analysis of the programmes underlying educational theory and organizational features, the contributions of health care professionals from the multiprofessional health centres and intervening partners, the link with the hospital, the link with local players, particularly medico-social players, and the patients participating in the programme.

SECONDARY OUTCOMES:
Number of Health care programmes developed in multiprofessional health centres realised in France | 7 months
Number of Health care programmes developed in multiprofessional health centres realised each year since 2014 in France | 7 months
Number of Health care programmes developed in multiprofessional health centres realised in each health authority agency | 7 months
Descriptive data of self-management programmes' characteristics developed in multiprofessional health centres, since 2014 | 7 months
  Number and percentage of programmes according to the coordinator's profession, Average number of multiprofessional health centres involved in each self-management programmes and percentage of self-management programmes according to the professions involved, Number and percentage of self-management programmes with co-construction with a patient association, Average number of years of existence of the self-management programmes initiated by multiprofessional health centres, Number and percentage of self-management programmes classified by theme, Number and percentage of self-management programmes by location (urban, semi-rural, rural), Number and percentage of renewal of self-management programmes among those in place for more than 4 years.
Self-management programmes characteristics associated with the continuation of self-management programmes in France | 7 months
  Type of health care professional, number of health care professional

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers

REFERENCES:
- [Result] Odgers-Jewell K, Ball LE, Kelly JT, Isenring EA, Reidlinger DP, Thomas R. Effectiveness of group-based self-management education for individuals with Type 2 diabetes: a systematic review with meta-analyses and meta-regression. Diabet Med. 2017 Aug;34(8):1027-1039. doi: 10.1111/dme.13340. Epub 2017 Mar 20. PMID 28226200
- [Result] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Result] Horigan G, Davies M, Findlay-White F, Chaney D, Coates V. Reasons why patients referred to diabetes education programmes choose not to attend: a systematic review. Diabet Med. 2017 Jan;34(1):14-26. doi: 10.1111/dme.13120. Epub 2016 Apr 15. PMID 26996982
- [Result] Mc Sharry J, Dinneen SF, Humphreys M, O'Donnell M, O'Hara MC, Smith SM, Winkley K, Byrne M. Barriers and facilitators to attendance at Type 2 diabetes structured education programmes: a qualitative study of educators and attendees. Diabet Med. 2019 Jan;36(1):70-79. doi: 10.1111/dme.13805. Epub 2018 Sep 21. PMID 30156335